CLINICAL TRIAL: NCT01889277
Title: A Phase II, Randomised, Double-blind, Placebo-controlled Study of MT-3995 in Subjects With Diabetic Nephropathy
Brief Title: Safety, Tolerability and Pharmacokinetic Study of MT-3995 in Subjects With Diabetic Nephropathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MT-3995-J03
Record Dates: First submitted 2013-06-26; First posted 2013-06-28 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Diabetic Nephropathy
Keywords: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- MT-3995-Low (Experimental): MT-3995-Low Dose
  Interventions: Drug: MT-3995-Low
- MT-3995-High (Experimental): MT-3995-High Dose
  Interventions: Drug: MT-3995-High
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT-3995-Low
  Arms: MT-3995-Low
Drug: MT-3995-High
  Arms: MT-3995-High
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate safety, tolerability and pharmacokinetics of MT-3995 in Subjects with Diabetic Nephropathy

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Type 2 diabetes mellitus and diabetic nephropathy, who have been treated with a stable dose of angiotensin converting enzyme-inhibitor (ACE-I) or angiotensin II receptor blocker (ARB)
* Glycosylated haemoglobin (HbA1c) ≤10.5%
* Subject with albuminuria

Exclusion Criteria:

* History of Type 1 diabetes, pancreas or β-cell transplantation, or diabetes secondary to pancreatitis or pancreatectomy.
* Serum potassium level <3.5 or >5.0 mmol/L
* Subjects who had acute kidney injury within 3 months prior to baseline or have undergone hemodialysis at any time prior to randomisation
* Subjects with clinically significant hypotension

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Frequency and nature of treatment-emergent adverse events and serious adverse events. | 20 weeks
Plasma concentrations of MT-3995 and its major metabolite | 20 weeks

SECONDARY OUTCOMES:
Change from baseline in Urine albumin-to-creatinine ratio (UACR) and blood pressure | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Masaomi Nangaku, Professor, Study Director — Division of Nephrology and Endocrinology University of Tokyo School of medicine; Kazuoki Kondou, Adviser, Study Director — Tanabe Pharma Corporation
Locations (1):
- Koukan Hospital, Kawasaki, Kanagawa Pref., Japan